CLINICAL TRIAL: NCT06461325
Title: Surgical Management Of Gastroschisis With Analysis Of Health Costs And Satisfaction Questionnaire On The Quality Of The Scar: A Retrospective Single-Center Comparative Study
Brief Title: Surgical Management Of Gastroschisis
Acronym: LAPS
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-CF-264
Record Dates: First submitted 2024-06-05; First posted 2024-06-17 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-05

CONDITIONS: Gastroschisis; Neonatal Disease; Hernia, Umbilical; Complication,Postoperative
Keywords: Gastroschisis; Hospitalization Costs; Neonate; Management
MeSH Terms: conditions — Gastroschisis; Infant, Newborn, Diseases; Hernia, Umbilical; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Bianchi: Gastroschisis treated by the Bianchi procedure
- Schuster: Gastroschisis treated by the Schuster procedure
- Sutureless: Gastroschisis treated by the Sutureless procedure
- Vacuum Assisted Closure: Gastroschisis treated by Vacuum Assisted Closure

SUMMARY:
The investigators aim to analyze the management of children born with gastroschisis between January 2009 and December 2023, i.e. to evaluate post-operative follow-up, hospitalization costs, the risk of post-operative umbilical hernia, and the parents' and the child's appreciation of the scar.

DETAILED DESCRIPTION:
Gastroschisis is an abdominal wall anomaly that affects 3 in 10,000 live births, and in over 90% of cases is diagnosed before birth. In fetuses with gastroschisis, the intestine protrudes through a defect in the abdominal wall, usually to the right of the umbilical cord. Although the survival rate of live newborns with gastroschisis is over 90%, the risk of intrauterine fetal death is still 7.5 times higher than in the normal population, and gastroschisis can cause significant morbidity during the neonatal period.

The scientific literature suggests multiple options for each stage in the care of children with gastroschisis, both pre- and postnatally. Heterogeneity of practice exists even within the same geographical area, and deserves to be analyzed.

In this context, the investigators wish to analyze the management of children born with gastroschisis between January 2009 and December 2023, i.e. to evaluate post-operative follow-up, hospitalization costs, the risk of post-operative umbilical hernia, and the parents' and the child's appreciation of the scar.

ELIGIBILITY:
Inclusion Criteria:

* Patients born with gastroschisis between January 2009 and December 2023

Exclusion Criteria:

* Patients born with gastroschisis before January 2009 or after December 2023 Patients without gastroschisis

Ages: 1 Minute to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients born with gastroschisis between January 2009 and December 2023
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with medical complications | through study completion, an average of 1 year
  sepsis, infections,
Number of patients with surgical complications | through study completion, an average of 1 year
  disunion, hernia scar

SECONDARY OUTCOMES:
Length of stay | through study completion, an average of 1 year
  Length of stay
Rate of Hospitalization Cost by patient | through study completion, an average of 1 year
  Costs by department, overall costs

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Destinval, Study Director — University Hospital, Clermont-Ferrand
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, Auvergne, France